CLINICAL TRIAL: NCT06787456
Title: Establishment of "Xijiang Project" Million-Person Screening Cohort for Nasopharyngeal Carcinoma
Brief Title: "Xijiang Project" Screening Cohort for NPC
Status: Active, not recruiting | Type: Observational
Sponsor: Ming-Yuan Chen (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chen, Professior, Chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: ZDWY.BYAFZZX.030
Record Dates: First submitted 2025-01-02; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma (NPC); Screening
Keywords: Nasopharyngeal Carcinoma (NPC); screening; Epstein-Barr virus; EBV DNA; EBV antibody
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — nasopharyngeal brushing, saliva, peripheral blood, etc.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening cohort of nasopharyngeal carcinoma: Population participating in nasopharyngeal carcinoma screening, aged between 30 and 69 years old.
  Interventions: Diagnostic Test: EBV antibodies test; Diagnostic Test: EBV DNA test; Other: epidemiological information survey; Other: Clinical examinations for high-risk participants; Other: EBV and human genetic sequencing

INTERVENTIONS:
Diagnostic Test: EBV antibodies test — ELISA test of VCA-IgA, EBNA1-IgA, EA-IgA, Zta-IgA, Rta-IgG and P85-Ab in nasopharyngeal brushing and plasma in plasma, saliva and nasopharyngeal brushing.
Diagnostic Test: EBV DNA test — quantitative polymerase chain reaction, methylation sequencing and target sequencing of EBV DNA in nasopharyngeal brushing, saliva and plasma.
Other: epidemiological information survey — epidemiological information survey including basic conditions, dietary and lifestyle habits, social, geographical, environmental, and other information.
Other: Clinical examinations for high-risk participants — nasopharyngoscopy, head and neck MRI.
Other: EBV and human genetic sequencing — EB virus and human genetic sequencing for plasma, etc.

SUMMARY:
The purpose of this study is to establish a comprehensive and integrated nasopharyngeal carcinoma screening cohort, which includes an epidemiological information database containing basic information, gender, age, ethnic and family history, dietary and lifestyle habits, and geographical environmental factors; a biobank of blood, tissue fluid, swabs, etc., for Epstein-Barr virus, tumors, and genetics; a clinical examination database including nasopharyngoscopy, imaging, pathology, and other examinations; and databases of Epstein-Barr virus and human genetic sequencing, etc.

DETAILED DESCRIPTION:
This study aims to initiate a multicenter prospective nasopharyngeal carcinoma (NPC) screening cohort study around China, starting from regions with high incidence of NPC, to conduct a million-person-scale screening cohort study. Participants who meet the selection criteria will be included in the cohort. All participants will undergo an epidemiological information survey (including basic conditions, dietary and lifestyle habits, social, geographical, environmental, and other information) through questionnaires, and various samples such as blood, tissue fluid, and throat swabs will be collected. Quantitative testing or genetic sequencing will be conducted on Epstein-Barr virus (EBV) (including EBV-related proteins, antibodies, EBV DNA quantification and sequence length, methylation levels, and next-generation sequencing), nasopharyngeal epithelial or tumor cells, etc., to establish, validate, optimize, and promote the optimal combination screening strategy for NPC; participants defined as high-risk of NPC by screening will undergo clinical nasopharyngoscopy and combined imaging and pathological examinations to confirm NPC patients and provide them with precise clinical treatment; regular follow-ups of the entire cohort will be conducted to study the risk factors and molecular mechanisms of NPC. The purpose of this study is to establish a comprehensive and integrated data platform, primarily based on the population from the South China, including an NPC epidemiological information database based on the gender, age, ethnicity, dietary and lifestyle habits, and geographical environmental factors, a biobank based on various samples and screening test results, and a clinical examination database based on nasopharyngoscopy, head and neck MRI, and a database for EB virus and human genetic sequencing information, etc., forming a multi-source heterogeneous, open, and shared data platform. Based on this data platform, basic scientific and clinical research on NPC will be conducted, including: developing, validating, and optimizing new NPC screening markers and their composite screening programs, clarifying the target population for the promotion of NPC composite screening programs; research study of the etiology and risk factors of NPC from genetic, ethnic, geographical, environmental, and lifestyle aspects, proposing a dynamic evolutionary molecular theory of NPC occurrence and development; exploring NPC prevention measures through lifestyle changes, vaccination interventions, and other methods; exploring new de-escalation clinical treatment plans for NPC, constructing new strategies for precise prevention and treatment of NPC such as minimally invasive surgical treatment and de-escalation of chemoradiotherapy, etc.

ELIGIBILITY:
Inclusion Criteria:

* Residents with a definite native place;
* Aged 30 and 69 years at screening;
* Capable of long-term cooperation with screening and follow-up.

Exclusion Criteria:

* Known severe cardiovascular, liver or kidney disease, or neuropsychiatric disorders;
* History of previous malignant tumors;
* Severe autoimmune diseases or immunodeficiency;
* Females with a positive pregnancy test at screening;
* Inability to cooperate with the study due to psychological, social, family, and geographical reasons.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents with a definite native place, aged 30 and 69 years at screening, and capable of long-term cooperation with screening and follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
A data platform for an NPC screening cohort | At screening, 3 years and 10 years thereafter
  A data platform, including an NPC epidemiological information database based on the gender, age, ethnicity, dietary and lifestyle habits, and geographical environmental factors, a biobank based on various samples and screening test results, and a clinical examination database based on nasopharyngoscopy, head and neck MRI, and a database for EB virus and human genetic sequencing information.

SECONDARY OUTCOMES:
Prevalence and incidence rate of nasopharyngeal carcinoma | At screening, 3 years and 10 years thereafter
  Endoscopy combined with or without biopsy is performed to evaluate the prevalence and rate of new cases of nasopharyngeal carcinoma, in a cohort study, and to identify the associated factors related with nasopharyngeal carcinoma.
Nasopharyngeal Carcinoma Death Rates | At screening, 3 years and 10 years thereafter
  Nasopharyngeal Carcinoma deaths confirmed in participants by a death review committee if available, otherwise by death certificate. Rate is the number of deaths divided by person years of follow-up in the study.
Death Rates From All Causes | At screening, 3 years and 10 years thereafter
  Deaths confirmed in participants by a death review committee if available, otherwise by death certificate. Rate is the number of deaths divided by person years of follow-up in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-yuan Chen, MD, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China